CLINICAL TRIAL: NCT03987880
Title: Comparison of a 4-mm Ring Shaped and 3.5-mm Ring Shaped PiXL Protocol for Low Grade Myopia
Brief Title: Photorefractive Intrastromal Corneal Crosslinking as a Treatment for Low Grade Myopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: Glaukos Corporation (Industry)
Responsible Party: Principal Investigator, Anders Behndig, Principal Investigator, Umeå University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PiXLMYOP-II
Record Dates: First submitted 2019-06-12; First posted 2019-06-17 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Myopia; Corneal Crosslinking; Refractive Errors; Eye Diseases
MeSH Terms: conditions — Myopia; Refractive Errors; Eye Diseases | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Prospective, single-masked intraindividually comparing randomized controlled trial. Participants will be randomized to receive ultraviolet (UV) light according to protocol A in one eye and protocol B in the other, which is masked to the participant. Both eyes will be treated during the same visit. Participants are randomized utilizing a computer list of unique random numbers between 1 and 27; an even number will be treated with the 4.0-mm zone in the right eye; an uneven number with the 4.0-mm zone in the left eye.
Who Masked: Participant
Masking Description: The participants are not aware which eye will receive the 4.0-mm ring-shaped zone treatment and which eye will receive the 3.5-mm ring-shaped zone treatment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 4.0 mm zone (Active Comparator): PiXL treatment with UV irradiation in a central 4.0-mm ring-shaped zone of the cornea. The area consist of three rings with a central 2-mm zone that is left untreated. The energy is higher towards the periphery of the ring-shaped area, reaching its maximum at 2-mm from the corneal centre. Pulsed UV-light, 1s on / 1s off; 30mW. For myopia of less than 0.75D, 10 J/cm2 is used, for higher levels of myopia 15J/cm2 is used.
  Interventions: Procedure: 4.0 mm treatment
- 3.5 mm zone (Experimental): PiXL treatment with UV irradiation in a central ring-shaped 3.5-mm zone of the cornea, with a central 1.5 mm zone that is left untreated. The illumination area consists of three rings, where the outer and inner ring are thinner than the middle ring. The maximum energy is distributed in the middle ring. Pulsed UV-light, 0.5s on / 1s off; 45mW. For myopia of less than 0.75D, a maximum of 10 J/cm2 is used, for higher levels of myopia a maximum of 15J/cm2 is used.
  Interventions: Procedure: 3.5 mm treatment

INTERVENTIONS:
Procedure: 4.0 mm treatment — PiXL treatment with UV irradiation in a central 4.0-mm ring-shaped zone of the cornea.
  Arms: 4.0 mm zone
Procedure: 3.5 mm treatment — PiXL treatment with UV irradiation in a central 3.5-mm ring-shaped zone of the cornea.
  Arms: 3.5 mm zone

SUMMARY:
To assess the improvement in refractive error and the corneal endothelial safety with a customized corneal crosslinking treatment regimen for low grade myopia. The study compares two treatment protocols, a 4.0-mm central ring-shaped zone with a 3.5-mm central ring-shaped zone in high oxygen environment without corneal epithelial debridement.

DETAILED DESCRIPTION:
The study design is a prospective, single-masked intraindividually comparing randomized controlled trial, conducted at the Department of Clinical Sciences / Ophthalmology, Umeå University Hospital, Umeå, Sweden. The study includes healthy men and women with low grade myopia, aged between 18-35 years and involves 27 participants with a myopia of -0.5 to -2.5 diopters (D) and astigmatism of ≤0.75D. All participants are treated with phototherapeutic intrastromal corneal collagen cross-linking (PiXL) without epithelial debridement (epi-on), after topical riboflavin. Both eyes are treated and randomized to receive ultraviolet (UV) light according to PiXL 4.0 mm treatment zone in one eye and PiXL 3.5 mm treatment zone in the other, which is masked to the participant. For myopia <0.75D, 10 J/cm^2 is used and for higher levels of myopia 15J/cm^2 is used. Throughout the treatment, humidified oxygen is continuously delivered around the eye using an oxygen mask to achieve an oxygen concentration of ≥95 percentage. All participants are informed about the procedures and provide oral and written consent before inclusion in the study.

At baseline, each eye is examined with slit-lamp microscopy, subjective refraction, determination of uncorrected (UCVA), low contrast visual acuity at 2.5 percentage and 10 percentage contrast and best corrected (BSCVA) visual acuities using the LogMAR fast protocol and intraocular pressure (IOP) using Goldmann applanation tonometry. Under standardized, mesopic light conditions each eye is evaluated by keratometry readings, central corneal thickness and after treatment also the depth of demarcation lines, extracted from Schemipflug camera measurements, Pentacam HR® (Oculus, Inc. Lynnwood, WA). Central corneal endothelial photographs are taken with the Topcon SP-2000P specular microscope (Topcon Europe B.V., Capelle a/d Ijssel, the Netherlands), from which the corneal endothelial cell count is manually calculated from a cluster of 25 cells from each photograph. Total ocular wavefront is measured with iTrace (Tracey Technologies, Inc.).

All the above mentioned examinations are reassessed at 1, 3 and 6 and 12 months after treatment. At 1 day and 1 week after treatment, solely UCVA, Auto refractor measurements, slit-lamp examination and a subjective comparison of discomfort and visual performance in each eye are evaluated.

ELIGIBILITY:
Inclusion Criteria:

Spherical equivalent on distance subjective refraction between -0.50D and -2.50D.

* Astigmatism ≤ 0.75D
* Stable myopia. Maximum change in refraction of 0.50D in the last 2 years.
* Best corrected visual acuity of at least 0.00 logMAR (ETDRS chart).
* Thinnest pachymetry reading ≥ 440 μm.
* No previous ocular surgery.
* No cognitive insufficiency interfering with the informed consent.

Exclusion Criteria:

* History of or current condition, disease, surgery or medication with ocular effects that could affect the outcomes of the treatment.
* Allergy to any substance or device used in the study.
* Cognitive insufficiency interfering with the informed consent.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline in uncorrected visual acuity | 1, 3, 6, 12 and 24 months after treatment
  Change from baseline in distance uncorrected visual acuity
Change from baseline in spherical equivalent | 1, 3, 6, 12 and 24 months after treatment
  Change from baseline in spherical equivalent on subjective distance refraction

SECONDARY OUTCOMES:
Change from baseline in corneal endothelial cell density | 12 and 24 months after treatment
  Change from baseline in central corneal endothelial cell density
Change from baseline in best corrected visual acuity | 1, 3, 6, 12 and 24 months after treatment
  Change from baseline in best spectacle corrected distance visual acuity

CONTACTS AND LOCATIONS:
Overall Officials: Anders Behndig, MD, PhD, Principal Investigator — Department of Clinical Sciences/Ophthalmology, Umeå University, Umeå, Sweden
Locations (1):
- Department of Clinical Sciences/Ophthalmology, Umeå University, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: No